CLINICAL TRIAL: NCT03451955
Title: The Effect of a Gluten Free Diet on the Permeability of the Blood Brain Barrier in Patients With Clinically Isolated Syndrome Measured by Dynamic Contrast Enhanced Magnetic Resonance Imaging
Brief Title: The Effect of a Gluten Free Diet on the Permeability of the Blood Brain Barrier in Patients With CIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Jens Rikardt Andersen, Associate professor, University of Copenhagen
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-17019986
Record Dates: First submitted 2017-09-22; First posted 2018-03-02 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Optic Neuritis; Multiple Sclerosis; Clinically Isolated Syndrome
Keywords: gluten; gluten free diet; blood brain barrier permeability; intestinal permeability; neuroinflammation; autoimmunity
MeSH Terms: conditions — Optic Neuritis; Multiple Sclerosis; Neuroinflammatory Diseases; Autoimmune Diseases | interventions — Diet, Gluten-Free

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients in the intervention group follow a gluten-free diet for six months.
  Interventions: Other: Gluten-free diet
- Control group (No Intervention): Patients in the control group follow their usual diet for six months

INTERVENTIONS:
Other: Gluten-free diet — Participants in the intervention group abstain from gluten for 6 months.
  Arms: Intervention group

SUMMARY:
Disruption of the blood brain barrier (BBB) is associated with inflammatory conditions of the central nervous system (CNS). This clinical trial aims to investigate whether following a gluten-free diet (GFD) for six months can contribute to normalizing BBB permeability in patients with newly diagnosed clinically isolated syndrome (CIS) and multiple sclerosis (MS). Furthermore, the study seeks to identify possible effects of a GFD on markers of systemic as well as CNS inflammation. Lastly, gut permeability is measured in order to examine whether there are any correlations between the permeability of the gut and the BBB as well as the inflammatory state in the intestine and CNS. From a patient's view, potential positive effects of a GFD will be manifested through an alleviation of symptoms, improved quality of life and reduced risk of CIS progressing to MS. Evaluating a possible role of gluten in MS pathogenesis can contribute to directing future research and optimizing treatment protocols.

DETAILED DESCRIPTION:
Background:

Disruption of the blood brain barrier (BBB) is believed to play a critical role in the pathogenesis of multiple sclerosis (MS). Cramer et al. (2014) found increased BBB permeability in MS patients compared to healthy controls (HC) with values being higher in cases with recent relapses (1). Furthermore, BBB permeability can contribute to predicting the conversion of optic neuritis (ON) to MS (2). In the same study, significant correlations were found between BBB permeability, leukocyte counts and levels of the chemokine CXCL10 in cerebrospinal fluid (CSF). Chemokines are believed to contribute to MS pathogenesis by attracting leukocyte populations to the CNS.

Sørensen et al. (1999) found elevated levels of the cytokines CXCL9, CXCL10 and CCL5 together with their receptors CXCR3 and CCR5 on leukocytes in CSF from MS patients during attacks (3). CXCR3 is expressed in human enterocytes, endothelial cells in the BBB and a variety of immune cells. Elevated expression of CXCR3 has also been measured on T cells from MS patients compared to HC, and in patients during relapses compared to remission (4). Exposure of intestinal epithelial cell lines to gliadin has been shown to activate the chemokine receptor CXCR3 and hereby leading to release of zonulin (5). Ex vivo experiments illustrated that zonulin, which has been identified as pre-haptoglobin 2, leads to a time- and dose dependent, reversible reduction of the transepithelial electrical resistance (TEER) of murine small intestinal mucosa (6). The effects of zonulin on gut permeability are assumed to be due to disruption of tight junctional integrity.

A pilot study (7) showed a higher proportion of individuals with increased intestinal permeability among patients with MS compared to sex-matched HC. A randomized clinical trial showed beneficial effects of a gluten-free diet (GFD) on annual relapse rate, lesional activity and expanded disability status scale (EDSS) in patients with relapsing-remitting MS (RRMS), when compared to a regular diet (8). Additionally, findings of significantly higher titers of IgA against gliadin, gluten and casein in MS patients compared to HC, could indicate a role of nutritional factors in MS (8).

The role of gluten in the pathogenesis of celiac disease (CD) is established. In CD dietary intake of gluten leads to the development of autoantibodies against the enzyme transglutaminase 2 (TG2). White matter autopsies have shown TG2 immunoreactivity in astrocytes from activated MS lesions (9). Furthermore, treatment with TG2 inhibitors led to attenuation of demyelination and clinical deficits in rats with chronic-relapsing experimental autoimmune encephalomyelitis (EAE) (10). A GFD has also been documented to protect against type 1 diabetes (T1D) in mice (11) and prolong the asymptomatic period after diagnosis of T1D in humans (12).

Lastly, gliadin fragments have been documented to stimulate the production of TNF-α and IL-8 in human monocytes directly (13). TNF-α has also been shown to have a regulatory effect on zonulin and to increase the permeability of the endothelial and epithelial cell layers (14), which could be an indirect mechanism through which gluten can induce alterations of gut and possibly also BBB permeability. A high gluten intake could thereby not only increase the influx of antigens, but also activate pathways of the innate immune system. This can theoretically contribute to establishing an inflammatory milieu and thereby facilitate the activation of autoreactive T cells. It could be hypothesized that the role of gluten in autoimmunity is not restricted to gluten itself being recognized as an antigen by people with specific HLA genotypes, but gluten might also increase the risk of losing tolerance against other antigens.

Purpose:

The study aims to investigate whether a GFD can contribute to decreasing BBB permeability in patients with ON, other clinically isolated syndrome (CIS) and MS. Furthermore, the study seeks to identify possible effects of a GFD on markers of systemic as well as CNS inflammation. Lastly, gut permeability is measured in order to examine whether there are any correlations between the permeability of the gut and the BBB as well as the inflammatory state in the intestine and CNS. Evaluating the effects of gluten intake on disease progression could contribute to identifying crucial mechanisms that underlie the pathogenesis of CIS and MS, directing future research and designing new, optimized treatment protocols.

Hypothesis:

Gluten may increase intestinal permeability and thereby elevate antigen influx possibly by activating CXCR3 on enterocytes. Increased gut permeability, gut inflammation and absorption of larger gliadin molecules may be associated with increased permeability of the BBB. Activation of BBB endothelial cells may lead to loss of tight junctional integrity, but also increased integrin expression and thereby enhanced extravasation of immune cells into the CNS.

Expected research value:

The study can contribute to a better understanding of the pathologies of ON and MS and provide a basis for the development of new treatment protocols. Conducting evidence-based research regarding the possible effects of gluten intake on the progression of autoimmune diseases will reduce misinformation as well as shed light on practical challenges associated with the implementation of dietary interventions for treatment purposes. The study is approved of the Scientific Ethics Committee.

Methods:

The trial is a clinically controlled, open label, intervention study including 40 patients with newly diagnosed CIS or MS. Patients will be divided into an intervention group and a control group, each of 20 patients. The intervention group will abstain from gluten for six months, while patients in the control group will retain their usual dietary habits. Before and after the intervention period, a variety of measurements will be conducted. These include:

* Anthropometric measurements: conducted to monitor possible effects of the GFD on participants´ body composition.
* Diet and lifestyle surveys: used to monitor participants´ dietary habits, smoking status, exercise, physical activity, sleeping pattern and quality of life.
* Clinical measures: Relapses, expanded disability status scale (EDSS), MS diagnosis, disease modifying treatment, T2 lesions count and lesion load. Treatment status and recent relapses will be used as covariates in the logistic regression analysis.
* Dynamic contrast-enhanced MRI: used to measure the permeability of the BBB in several tissue subtypes (normal appearing white matter and grey matter and MS lesions) as segmented on high resolution T2 FLAIR and 3D T1 weighted images. The number of new or enhancing lesions is being monitored.
* Intestinal permeability test: conducted to measure intestinal permeability and absorption capacity.
* Lumbar puncture: used to determine disease activity in the CNS. Analyses include pre-haptoglobin 2, oligoclonal bands, TNF-α, IL-1β, IL-8, INF-γ, CXCL9, CXCL10, CCL5, immune cell counts, expression of CXCR3 on immune cells.
* Blood samples: used to determine the grade of inflammation outside the CNS and diagnose celiac disease. Analyses include S100β, pre-haptoglobin 2, anti-gliadin antibodies, CRP, TNF-α, IL-1β, INF-γ, immune cell counts, expression of CXCR3 on immune cells, endotoxin, intestinal fatty acid binding protein, 25-(OH)-cholecalciferol.
* Fecal samples: used to measure gut microbiota profiling and short chain fatty acids.

BBB and intestinal permeability will not only be measured through an MRI scan and an intestinal permeability test respectively, but also using the biomarker zonulin. Of notice is that our measurements of zonulin in CSF (for BBB permeability) and serum (for intestinal permeability) will be carried out in collaboration with Assistant Professor Dr. Ian Galea, who has established a unique analytical method, based on western blotting using a non-commercially, proprietary antibody manufactured by Biorad, for this purpose. Every other assay used in the scientific community measures both haptoglobin and zonulin, whereas our assay measures only zonulin and is therefore characterized by increased accuracy.

Expected results:

A gluten-free diet is expected to alleviate CIS symptoms, improve quality of life and reduce the risk of CIS progressing into MS. Mechanistically this is expected to be manifested through a normalized BBB and intestinal permeability, decreased lesional activity and by dampening the activity of a previously overactive immune system. If our hypothesis is proven to be correct, MS and CIS patients should be informed about the results of the study and the option of following a GFD could potentially become part of the standardized patient treatment in hospitals.

Publication of results:

Results will be published independent of study outcome. Positive, negative as well as inconclusive results will be published. Results are expected to be published in peer-reviewed international journals.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women ≥18 and ≤59 years of age
* Patients with newly diagnosed CIS or MS deemed physically and mentally able to participate in a study

Exclusion Criteria:

* More conflicting disorders in the same patient
* Pregnancy and lactating women and women planning pregnancy during the study period
* People with severe claustrophobia
* People with MR incompatible implants/ foreign objects, including implanted pacemakers, heart valve prostheses, prostheses in the middle ear, implanted devices (e.g. insulin pump), metal debris, e.g. metal splinters in the eyes, miscellaneous shunts and catheters, metal clips from operations
* Surgeries within the last 6 weeks
* Previous reactions to MR contrast agent, bronchial asthma or history of other allergies
* Elevated serum creatinine
* People already on a gluten restricted/ GFD

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
Permeability of the blood brain barrier | Change from baseline at 6 months
  Blood brain barrier permeability measured by contrast enhanced magnetic resonance imaging as well as concentration of pre-haptoglobin 2 in CSF

SECONDARY OUTCOMES:
Intestinal permeability | Change from baseline at 6 months
  Measured by lactulose/mannitol intestinal permeability test and concentration of pre-haptoglobin 2 in blood
Intestinal absorption capacity | Change from baseline at 6 months
  Measured by D-xylose test
Counts of T cell subpopulations in peripheral blood and CSF | Change from baseline at 6 months
  Flow cytometry analysis using antibodies for CD3, CD8, CD4, CD45RA, CXCR3, CCR6, CCR4, CCR9, integrins alpha4, beta7 and beta1
Macrophage activation in peripheral blood and CSF | Change from baseline at 6 months
  Soluble CD163 in peripheral blood and CSF measured by ELISA
Neuroinflammation | Change from baseline at 6 months
  Measured as neurofilament light chain in CSF and peripheral blood
Bacterial translocation | Change from baseline at 6 months
  Measured as endotoxin in blood by ELISA
Osteopontin as a marker of disease activity in multiple sclerosis | Change from baseline at 6 months
  Measured in blood and CSF by ELISA
Enterocyte damage | Change from baseline at 6 months
  Measured as intestinal fatty acid binding protein in blood by ELISA
Gut microbiota profiling | Change from baseline at 6 months
  Measured in feces by 16S rRNA sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Jens Rikardt Andersen, Study Director — University of Copenhagen
Locations (2):
- Denmark (2):
  - University of Copenhagen, Copenhagen, Frederiksberg
  - Rigshopitalet, Glostrup Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cramer SP, Simonsen H, Frederiksen JL, Rostrup E, Larsson HB. Abnormal blood-brain barrier permeability in normal appearing white matter in multiple sclerosis investigated by MRI. Neuroimage Clin. 2013 Dec 10;4:182-9. doi: 10.1016/j.nicl.2013.12.001. eCollection 2014. PMID 24371801
- [Background] Cramer SP, Modvig S, Simonsen HJ, Frederiksen JL, Larsson HB. Permeability of the blood-brain barrier predicts conversion from optic neuritis to multiple sclerosis. Brain. 2015 Sep;138(Pt 9):2571-83. doi: 10.1093/brain/awv203. Epub 2015 Jul 17. PMID 26187333
- [Background] Sorensen TL, Tani M, Jensen J, Pierce V, Lucchinetti C, Folcik VA, Qin S, Rottman J, Sellebjerg F, Strieter RM, Frederiksen JL, Ransohoff RM. Expression of specific chemokines and chemokine receptors in the central nervous system of multiple sclerosis patients. J Clin Invest. 1999 Mar;103(6):807-15. doi: 10.1172/JCI5150. PMID 10079101
- [Background] Andalib A, Doulabi H, Najafi M, Tazhibi M, Rezaie A. Expression of chemokine receptors on Th1/Th2 CD4+ lymphocytes in patients with multiple sclerosis. Iran J Immunol. 2011 Mar;8(1):1-10. PMID 21427490
- [Background] Lammers KM, Lu R, Brownley J, Lu B, Gerard C, Thomas K, Rallabhandi P, Shea-Donohue T, Tamiz A, Alkan S, Netzel-Arnett S, Antalis T, Vogel SN, Fasano A. Gliadin induces an increase in intestinal permeability and zonulin release by binding to the chemokine receptor CXCR3. Gastroenterology. 2008 Jul;135(1):194-204.e3. doi: 10.1053/j.gastro.2008.03.023. Epub 2008 Mar 21. PMID 18485912
- [Background] Tripathi A, Lammers KM, Goldblum S, Shea-Donohue T, Netzel-Arnett S, Buzza MS, Antalis TM, Vogel SN, Zhao A, Yang S, Arrietta MC, Meddings JB, Fasano A. Identification of human zonulin, a physiological modulator of tight junctions, as prehaptoglobin-2. Proc Natl Acad Sci U S A. 2009 Sep 29;106(39):16799-804. doi: 10.1073/pnas.0906773106. Epub 2009 Sep 15. PMID 19805376
- [Background] Buscarinu MC, Cerasoli B, Annibali V, Policano C, Lionetto L, Capi M, Mechelli R, Romano S, Fornasiero A, Mattei G, Piras E, Angelini DF, Battistini L, Simmaco M, Umeton R, Salvetti M, Ristori G. Altered intestinal permeability in patients with relapsing-remitting multiple sclerosis: A pilot study. Mult Scler. 2017 Mar;23(3):442-446. doi: 10.1177/1352458516652498. Epub 2016 Jul 11. PMID 27270497
- [Background] van Strien ME, Drukarch B, Bol JG, van der Valk P, van Horssen J, Gerritsen WH, Breve JJ, van Dam AM. Appearance of tissue transglutaminase in astrocytes in multiple sclerosis lesions: a role in cell adhesion and migration? Brain Pathol. 2011 Jan;21(1):44-54. doi: 10.1111/j.1750-3639.2010.00428.x. Epub 2010 Aug 20. PMID 20731658
- [Background] van Strien ME, de Vries HE, Chrobok NL, Bol JGJM, Breve JJP, van der Pol SMP, Kooij G, van Buul JD, Karpuj M, Steinman L, Wilhelmus MM, Sestito C, Drukarch B, Van Dam AM. Tissue Transglutaminase contributes to experimental multiple sclerosis pathogenesis and clinical outcome by promoting macrophage migration. Brain Behav Immun. 2015 Nov;50:141-154. doi: 10.1016/j.bbi.2015.06.023. Epub 2015 Jun 29. PMID 26133787
- [Background] Antvorskov JC, Josefsen K, Engkilde K, Funda DP, Buschard K. Dietary gluten and the development of type 1 diabetes. Diabetologia. 2014 Sep;57(9):1770-80. doi: 10.1007/s00125-014-3265-1. Epub 2014 May 29. PMID 24871322
- [Background] Svensson J, Sildorf SM, Pipper CB, Kyvsgaard JN, Bojstrup J, Pociot FM, Mortensen HB, Buschard K. Potential beneficial effects of a gluten-free diet in newly diagnosed children with type 1 diabetes: a pilot study. Springerplus. 2016 Jul 7;5(1):994. doi: 10.1186/s40064-016-2641-3. eCollection 2016. PMID 27398272
- [Background] Jelinkova L, Tuckova L, Cinova J, Flegelova Z, Tlaskalova-Hogenova H. Gliadin stimulates human monocytes to production of IL-8 and TNF-alpha through a mechanism involving NF-kappaB. FEBS Lett. 2004 Jul 30;571(1-3):81-5. doi: 10.1016/j.febslet.2004.06.057. PMID 15280021
- [Background] Nouri M, Bredberg A, Westrom B, Lavasani S. Intestinal barrier dysfunction develops at the onset of experimental autoimmune encephalomyelitis, and can be induced by adoptive transfer of auto-reactive T cells. PLoS One. 2014 Sep 3;9(9):e106335. doi: 10.1371/journal.pone.0106335. eCollection 2014. PMID 25184418